CLINICAL TRIAL: NCT02289508
Title: Diagnostic and Prognostic Role of USCOM in Adult Patients With Heart Failure-A Prospective Observational Study
Brief Title: Role of USCOM in Adult Patients With Heart Failure
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Cardiff and Vale University Health Board (Other Government); University Hospitals, Leicester (Other)
Responsible Party: Principal Investigator, Timothy H Rainer, Director & Professor, Chinese University of Hong Kong
Other Study IDs: 2014.464
Record Dates: First submitted 2014-11-06; First posted 2014-11-13 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Acute Decompensated Heart Failure; Congestive Heart Failure Compensated
Keywords: Heart Failure; Hemodynamics; Echocardiography; Diagnostic techniques and procedures; Ultrasonography; USCOM
MeSH Terms: conditions — Heart Failure | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 10ml venous blood will be collected through venipuncture. Blood will be centrifuged, plasma decanted, and stored pending B-type Natriuretic Peptide (BNP) measurements.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- acute decompensated heart failure: Patients who fulfill Framingham criteria will be classified as acute decompensated heart failure (adHF). For this study we define this as an acute change in symptoms and signs within the previous 24 hours. When symptoms gradually deteriorate between one day and one month, it is described as gradual decompensated heart failure (gdHF). Some patients may have both.
  Interventions: Device: Ultrasonic cardiac output monitor; Device: Echocardiography
- compensated heart failure: compensated heart failure (cHF) is defined as the existence of heart failure in the absence of any acute exacerbation but which may either include typical chronic symptoms and signs or may be asymptomatic but with evidence of cardiac dysfunction i.e. a reduced ejection fraction.
  Interventions: Device: Ultrasonic cardiac output monitor; Device: Echocardiography
- non-heart failure patients: Non-heart failure patients (nHFp) are a patient control group with suspected heart failure but who after further assessment are found not to meet the criteria. Such patients may subsequently be found to have COPD, anaemia, over transfusion. As the purpose of this study is to assess the potential value of USCOM parameters in the assessment of patients with possible heart failure in the clinical setting, it is important to include patients without heart failure.
  Interventions: Device: Ultrasonic cardiac output monitor; Device: Echocardiography
- healthy controls: Healthy controls are subjects with not acute or chronic illness.
  Interventions: Device: Ultrasonic cardiac output monitor

INTERVENTIONS:
Device: Ultrasonic cardiac output monitor — An Ultrasonic Cardiac Output Monitor, a non-invasive Doppler ultrasonography, is capable of measuring haemodynamic parameters non-invasively and appears to be simple and rapid to use, portable, relatively inexpensive and has less potential complications compared with the standard technique, pulmonary artery thermodilution (PATD). It has been compared favorably with a wide range of standard techniques, including PATD, with good interobserver reliability. USCOM may help on monitoring HF and suggesting proper treatment in order to reduce the mortality of adHF.
  Other Names: USCOM
Device: Echocardiography — 2D-echo is a conventional standard-of-care tool for non-invasive hemodynamic assessments in adults. The use of 2D-echo requires highly trained personnel, and assessments may take anywhere between 30-45 minutes. It is used to find out the ejection fraction and to compare the haemodynamic parameters with USCOM in this study.
  Other Names: Echo
  Groups: acute decompensated heart failure; compensated heart failure; non-heart failure patients

SUMMARY:
Objective:

The Ultrasonic Cardiac Output Monitor (USCOM) is a non-invasive, quantitative method for measuring and monitoring cardiovascular haemodynamic parameters in patients. The aims of this study are:

1. To investigate whether USCOM-derived haemodynamic parameters such as Cardiac output (CO), inotropy and oxygen delivery (DO2) have a role in the diagnosis of patients with a compensated heart failure syndrome (cHFS) or acute decompensated heart failure syndrome (adHFS)
2. To investigate whether USCOM-derived haemodynamic parameters such as CO, inotropy and DO2 correlate with heart failure staging, especially New York Heart Association (NYHA) class and American Heart Association (AHA) stage.
3. To investigate whether USCOM-derived haemodynamic parameters such as velocity time interval (vti), stroke volume (SV), CO, SV index (SVI), CO index (CI), inotropy and DO2 correlate with ejection fraction.
4. To investigate whether USCOM-derived haemodynamic variables may be used as prognostic indicators of 30-day, 6-month and 1-year Major Adverse Cardiac Events (MACE).
5. To evaluate the agreement between hemodynamic measurements obtained using the Ultrasonic Cardiac Output Monitor (USCOM®; USCOM Ltd., Sydney, Australia), and reference standards as determined by 2 Dimensional echocardiography (2D-echo) measurements in groups of haemodynamically stable and unstable adult patients.

Design:

This prospective observational cohort study will be conducted in the Prince of Wales Hospital in Hong Kong.

Setting and Subjects:

Patients will be screened and recruited from adult patients either scheduled for elective 2D-echo at a cardiology clinic at the Prince of Wales Hospital, or attending the emergency department at the Prince of Wales Hospital.

Interventions:

Haemodynamic measurements made using the USCOM and 2D-echo will be compared. In order to assess inter-observer variability, a second, blinded operator will repeated 15% of scans.

DETAILED DESCRIPTION:
Acute heart failure syndromes (aHFS) cause almost 1 million hospitalizations annually in the United States and are the leading cause of hospitalization in persons aged over 65 years. In 2003, inpatient management of aHFS cost an estimated $12.7 billion in the United States. In 2003, 12.5% of the population in Hong Kong were aged over 65, the third highest proportion of elderly among all countries, and it is postulated that by 2033, the proportion of the elderly in the population will increase to 25%. With the growing elderly population, and the increasing prevalence of hypertension and ischemic heart disease (the major causes of heart failure), heart failure has become a major health care issue globally. In western countries the incidence ranges from 1 to 10 cases/1000/year. Other studies suggest that heart failure is a large and growing public health burden throughout Europe.

Acute exacerbation of heart failure symptoms is a common emergency department (ED) presentation and is known as acute decompensated heart failure (adHF). Acute decompensated heart failure represents the single greatest cost to the US hospitals funded by Medicaid. In Hong Kong (HK), the incidence rate of heart failure was 3-3.8/1000/year rising to 20/1000/year in women over the age of 85 years in recent years. It has been estimated that 7% of all acute medical admissions was due to this condition. In recent years there has been a 10% annual increase in admissions for patients with adHF. Currently in Hong Kong, the vast majority of ED patients with adHF are admitted as inpatients to hospital. In 2005, an audit of outcomes in patients with acute cardiogenic pulmonary oedema, the most severe manifestation of heart failure, presenting to the emergency department at the Prince of Wales Hospital showed that nearly 30% of patients die within 30 days, and a further 30% require readmission within 30 days. Recent evidence from the USA suggests that ED operated observation units are effective in managing low to medium risk adHF patients, reducing length of stay (LOS) for these patients without adversely affecting readmission rate, morbidity and mortality.

2 Dimensional echocardiography (2D-echo) is a conventional standard-of-care tool for non-invasive hemodynamic assessments in adults. In stable settings, heart failure is often characterized and classified according to ejection fraction measured by echocardiography which may be considered a pragmatic gold standard. However, the use of 2D-echo requires highly trained personnel. Obtaining measurements and calculating fundamental cardiovascular parameters such as cardiac output (CO)may take anywhere between 30 to 45 minutes, which is impractical for any setting, let alone an acute care setting. Further, such personnel are frequently not available in emergency departments. The feasibility of real time haemodynamic assessments is therefore limited with 2D-echo. More sophisticated echocardiographic techniques have been developed in an attempt to overcome the problems of sensitivity to preload and particularly afterload, but have achieved little penetration in critical care.

In acute critical care settings, the diagnosis of adHF is based on the history and clinical signs, sometimes aided by echocardiography, chest radiography and blood markers such as B-type Natriuretic Peptide (BNP). The value of BNP over clinical assessment in patients presenting with dyspnoea has been questioned and there is a need for other tools to improve diagnosis. Commencement, dosing, and withdrawal of vasopressors, vasodilators, and inotropes is still largely based on clinical assessment, sometimes assisted by measurement of surrogates of inotropy such as ejection fraction (EF) or aortic ejection velocity, despite the well-known shortcomings of these indices in critical care. This is particularly so in complex surgical patients where vascular tone and fluid loading status are highly variable and changing.

Heart failure is an abnormality of cardiac structure or function leading to failure of the heart to deliver oxygen at a rate commensurate with the requirements of the metabolizing tissues, despite normal filling pressures (or only at the expense of increased filling pressures). The commonest causes are hypertension or ischemic heart disease. If this definition holds, then heart failure should be associated with some measure of reduction in inotropy or oxygen delivery. Until recently there was no simple non-invasive, bedside test that could aid the assessment of patients with heart failure. Whilst inotropy (or myocardial contractility) as a concept is well known to all clinicians, it is seldom thought of as a measurable quantity.

USCOM has been introduced as a non-invasive bedside haemodynamic monitoring tool that utilizes continuous-wave Doppler ultrasound. The USCOM has a number of advantages. It accuracy, validity and reasonable precision has been confirmed by many studies and in a variety of contexts. It is easily portable, takes only several minutes to obtain reliable measurements in most cases, and can be conducted by trained physicians or nurses.

Some studies have shown good agreement between USCOM and echocardiography but others have been less convincing. With this in mind, there is still a need for further studies to confirm or refute levels of agreement between USCOM and echocardiography.

The potential utility of USCOM for assessing patients with adHF has recently been suggested. Inotropy measurements derived from USCOM are greatly reduced in patients with New York Heart Association (NYHA) Class IV and American Heart association (AHA) stage C, acute left ventricular failure, when compared with healthy controls. These findings have led to the proposal that as USCOM can measure inotropy, then it could be used to assess and to manage heart failure. Although inotropy, derived by USCOM, is low in patients with adHF and NYHA class IV, nevertheless there is no evidence of a dose-relationship between USCOM-derived inotropy and NYHA class, or of a correlation with increasing severity of adHF, with ejection fraction.

Many, if not most, emergency departments throughout the world do not have 2D-echo available 24 hours a day, if at all. The value of BNP testing to improve outcomes has been questioned but even if used, it is frequently not available in many hospitals. As such the assessment and diagnosis of heart failure, and the means to monitor the effect of therapy, constitutes a major unmet need in clinical practice and especially in emergency departments.

Aim

The overall aim of this study is to investigate whether USCOM-derived haemodynamic parameters may have diagnostic, risk-stratification, prognostic and therapeutic monitoring potential in patients with suspected heart failure. The specific objectives are:

1. To investigate whether USCOM-derived haemodynamic parameters such as CO, inotropy and oxygen delivery (DO2) have a role in the diagnosis of patients with a compensated heart failure syndrome (cHFS) or acute decompensated heart failure syndrome (adHFS)
2. To investigate whether USCOM-derived haemodynamic parameters such as CO, inotropy and DO2 correlate with heart failure staging, especially NYHA class and AHA stage.
3. To investigate whether USCOM-derived haemodynamic parameters such as velocity time interval (vti), stroke volume (SV), CO, SV index (SVI), CO index (CI), inotropy and DO2 correlate with ejection fraction.
4. To investigate whether USCOM-derived haemodynamic variables may be used as prognostic indicators of 30-day, 6-month and 1-year Major Adverse Cardiac Events (MACE).
5. To evaluate the agreement between hemodynamic measurements obtained using the Ultrasonic Cardiac Output Monitor (USCOM®; USCOM Ltd., Sydney, Australia), and reference standards as determined by 2D-echo measurements in groups of haemodynamically stable and unstable adult patients.

Data collection and measurable parameters

* Demographics including sex, age, height and weight
* Chief complaints, concurrent illnesses and significant past history
* Clinical signs including respiration rate, heart rate, systolic blood pressure, diastolic blood pressure, oxygen saturation and CGS.
* USCOM derived haemodynamic parameters
* Full blood examination, urea and electrolytes, arterial or venous blood gases, blood glucose, lactate, BNP, ECG and chest x-ray
* ED diagnosis, disposition from ED, hospital length of stay, ICU length of stay, hospital diagnosis and in-hospital mortality All the above data will be entered into a database that is securely stored with access only by the investigators.

Definition of haemodynamic parameters:

* Flow time corrected (FTc) is calculated using Bazett's formula: FTc = FT/√tHR, where tHR = the heart beat period in seconds (s). The unit of FTc is ms.
* Velocity time integral (vti) is the integral of the flow profile, i.e. the distance the blood travels in one beat. The unit of vti is m/s.
* Cardiac output (CO) is the volume of blood pumped by the heart in one minute: CO = SV x HR. The unit is l/min.
* Cardiac index (CI) is equal to CO divided by BSA. The unit is l/min/m2.
* Inotropy index refers to (Potential energy + Kinetic energy) divided by body surface area. The unit of inotropy is W/m2.
* Minute distance (MD) is the distance a blood cell travels in metres per minute (m/min). MD = HR x vti, where vti = velocity time integral or stroke distance, which is the distance in centimetres (cm) a single reflector travels per cycle, and is defined as the area of the flow.
* Stroke volume (SV) is the volume of blood ejected from the heart during one systolic stroke. SV = vti x πr2,where πr2 = flow cross sectional area. The unit of SV is ml.
* Stroke volume index (SVI) is SV divided by BSA and the unit is ml/m2.
* Stroke volume variation (SVV) is the percentage change in SV between a group of beats. SVV = (SVmax - SVmin x 100) / [(SVmax + SVmin)/2].
* Systemic vascular resistance (SVR) is the pressure against which the heart pumps. SVR = MAP/CO. The unit is d.s.cm-5.
* Systemic vascular resistance index (SVRI) SVRI = SVR x BSA d.s.cm-5m2.
* Oxygen delivery (DO2) is calculated by the equation: DO2 = 1.34 x Hb x SpO2/100 x CO, where Hb = hemoglobin in grams of hemoglobin per litre of blood (g/l); SpO2 = the peripheral oxygen saturation as a percentage (%). The unit of DO2 is ml/min.
* Oxygen delivery index (DO2I) is equal to DO2 divided by BSA. The unit of DO2I is ml/min/m2.
* Inotropy index refers to (Potential energy + Kinetic energy) divided by body surface area. The unit of inotropy is W/m2.

This project will provide essential data on the potential for clinicians without access to echocardiography but with access to USCOM, to effectively and safely assess patients with cHF, and adHF. Confirming the value of USCOM will enable the earlier diagnosis of heart failure and cardiogenic shock, earlier appropriate management, will remove the guesswork and uncertainty as whether or not to administer diuretics, intravenous fluid, vasodilators, vasoconstrictors, inotropes, chronotropes or blockers. This will open the door for trials orientated to optimizing haemodynamics in the cold and acute critical care settings, thus permitting optimal use of life-saving therapies, and optimizing survival. Such early treatment options should reduce the need for admission to hospital and length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, AND
2. Written informed consent by patient or nearest relative where appropriate, AND Either
3. Referred for echocardiography, OR
4. At least one typical symptom and one typical sign consistent with possible heart failure, OR
5. Healthy volunteers

Exclusion Criteria:

* Age <18 years
* Prior enrollment in study
* Patients with known or suspected pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be screened and recruited from adult patients either scheduled for elective 2D-echo at a cardiology clinic at the Prince of Wales Hospital, or attending the emergency department at the Prince of Wales Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-02-06 (Actual); Study Completion 2018-02-06 (Actual)

PRIMARY OUTCOMES:
Difference in mean (SD) inotropy between New York Heart Association (NYHA) stages I, II, III and IV | On Day 1
  Inotropy = (Potential energy + kinetic energy) divided by BSA; measured at aortic and pulmonary window by USCOM; units W/m2

SECONDARY OUTCOMES:
Difference in mean (SD) vti, FTc, SV, SVI, CO, CI, MD, SVR, SVRI, SVV, DO2, DO2I, Inotropy and ejection fraction | On Day 1
  Please see an explanation of these variables and units in the section on detailed description
Difference in mean (SD) vti, FTc, SV, SVI, CO, CI, MD, SVR, SVRI, SVV, DO2, DO2I, Inotropy and AHA stage | On Day 1
  Please see an explanation in of these variables and units in the section on detailed description
Agreement between CO and SV measured separately by USCOM and 2D-Echo | On Day 1
  Cardiac output (CO) is the volume of blood pumped by the heart in one minute (CO = SV x HR); units L/min.
Number of subjects with and without Major Adverse Cardiac Events (MACE). | 30-days, 6-months and 1-year
  MACE are presented in total, and also as separate safety and intervention subgroups.
Number of subjects with and without acute decompensated heart failure syndrome (adHFS) | On Day 1
  The presence or absence of adHFS is defined according to the Framingham criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy H Rainer, MD FCEM, Principal Investigator — Accident & Emergency Medicine Academic Unit
Locations (1):
- Prince of Wales Hospital, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided
Data may be shared pending external requests.

REFERENCES:
- [Background] McMurray JJ, Stewart S. Epidemiology, aetiology, and prognosis of heart failure. Heart. 2000 May;83(5):596-602. doi: 10.1136/heart.83.5.596. No abstract available. PMID 10768918
- [Background] Mendez GF, Cowie MR. The epidemiological features of heart failure in developing countries: a review of the literature. Int J Cardiol. 2001 Sep-Oct;80(2-3):213-9. doi: 10.1016/s0167-5273(01)00497-1. PMID 11578717
- [Background] Sanderson JE, Tse TF. Heart failure: a global disease requiring a global response. Heart. 2003 Jun;89(6):585-6. doi: 10.1136/heart.89.6.585. No abstract available. PMID 12748201
- [Background] Hung YT, Cheung NT, Ip S, Fung H. Epidemiology of heart failure in Hong Kong, 1997. Hong Kong Med J. 2000 Jun;6(2):159-62. PMID 10895138
- [Background] Peacock WF. Acute Emergency Department management of heart failure. Heart Fail Rev. 2003 Oct;8(4):335-8. doi: 10.1023/a:1026187013370. PMID 14574053
- [Background] Peacock WF. Heart failure management in the emergency department observation unit. Prog Cardiovasc Dis. 2004 Mar-Apr;46(5):465-85. doi: 10.1016/j.pcad.2003.12.004. PMID 15179633
- [Background] Burkhardt J, Peacock WF, Emerman CL. Predictors of emergency department observation unit outcomes. Acad Emerg Med. 2005 Sep;12(9):869-74. doi: 10.1197/j.aem.2005.03.534. PMID 16141022
- [Background] Peacock WF. Using the emergency department clinical decision unit for acute decompensated heart failure. Cardiol Clin. 2005 Nov;23(4):569-88, viii. doi: 10.1016/j.ccl.2005.08.014. PMID 16278126
- [Background] Silver MA, Peacock WF 4th, Diercks DB. Optimizing treatment and outcomes in acute heart failure: beyond initial triage. Congest Heart Fail. 2006 May-Jun;12(3):137-45. doi: 10.1111/j.1527-5299.2006.05413.x. PMID 16760699
- [Background] Kosowsky JM, Gasaway MD, Hamilton CA, Storrow AB. Preliminary experience with an emergency department observation unit protocol for heart failure. Acad Emerg Med. 2000 Oct;7(10):1171. PMID 11015282
- [Background] Sanderson JE, Chan SK, Chan WW, Hung YT, Woo KS. The aetiology of heart failure in the Chinese population of Hong Kong--a prospective study of 730 consecutive patients. Int J Cardiol. 1995 Aug;51(1):29-35. doi: 10.1016/0167-5273(95)02398-g. PMID 8522394
- [Background] Diercks DB, Peacock WF, Kirk JD, Weber JE. ED patients with heart failure: identification of an observational unit-appropriate cohort. Am J Emerg Med. 2006 May;24(3):319-24. doi: 10.1016/j.ajem.2005.11.014. PMID 16635705
- [Background] Juan A, Salazar A, Alvarez A, Perez JR, Garcia L, Corbella X. Effectiveness and safety of an emergency department short-stay unit as an alternative to standard inpatient hospitalisation. Emerg Med J. 2006 Nov;23(11):833-7. doi: 10.1136/emj.2005.033647. PMID 17057132
- [Background] Kirkpatrick JN, Vannan MA, Narula J, Lang RM. Echocardiography in heart failure: applications, utility, and new horizons. J Am Coll Cardiol. 2007 Jul 31;50(5):381-96. doi: 10.1016/j.jacc.2007.03.048. Epub 2007 Jul 13. PMID 17662389
- [Background] Tei C, Ling LH, Hodge DO, Bailey KR, Oh JK, Rodeheffer RJ, Tajik AJ, Seward JB. New index of combined systolic and diastolic myocardial performance: a simple and reproducible measure of cardiac function--a study in normals and dilated cardiomyopathy. J Cardiol. 1995 Dec;26(6):357-66. PMID 8558414
- [Background] Kass DA, Maughan WL, Guo ZM, Kono A, Sunagawa K, Sagawa K. Comparative influence of load versus inotropic states on indexes of ventricular contractility: experimental and theoretical analysis based on pressure-volume relationships. Circulation. 1987 Dec;76(6):1422-36. doi: 10.1161/01.cir.76.6.1422. PMID 3454658
- [Background] Lam LL, Cameron PA, Schneider HG, Abramson MJ, Muller C, Krum H. Meta-analysis: effect of B-type natriuretic peptide testing on clinical outcomes in patients with acute dyspnea in the emergency setting. Ann Intern Med. 2010 Dec 7;153(11):728-35. doi: 10.7326/0003-4819-153-11-201012070-00006. PMID 21135296
- [Background] McMurray JJ, Adamopoulos S, Anker SD, Auricchio A, Bohm M, Dickstein K, Falk V, Filippatos G, Fonseca C, Gomez-Sanchez MA, Jaarsma T, Kober L, Lip GY, Maggioni AP, Parkhomenko A, Pieske BM, Popescu BA, Ronnevik PK, Rutten FH, Schwitter J, Seferovic P, Stepinska J, Trindade PT, Voors AA, Zannad F, Zeiher A; ESC Committee for Practice Guidelines. ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure 2012: The Task Force for the Diagnosis and Treatment of Acute and Chronic Heart Failure 2012 of the European Society of Cardiology. Developed in collaboration with the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2012 Jul;33(14):1787-847. doi: 10.1093/eurheartj/ehs104. Epub 2012 May 19. No abstract available. PMID 22611136
- [Background] Dey I, Sprivulis P. Emergency physicians can reliably assess emergency department patient cardiac output using the USCOM continuous wave Doppler cardiac output monitor. Emerg Med Australas. 2005 Jun;17(3):193-9. doi: 10.1111/j.1742-6723.2005.00722.x. PMID 15953218
- [Background] Patel N, Dodsworth M, Mills JF. Cardiac output measurement in newborn infants using the ultrasonic cardiac output monitor: an assessment of agreement with conventional echocardiography, repeatability and new user experience. Arch Dis Child Fetal Neonatal Ed. 2011 May;96(3):F206-11. doi: 10.1136/adc.2009.170704. Epub 2010 Jul 6. PMID 20605971
- [Background] Geiger S, Stemmler HJ, Suhl P, Stieber P, Lange V, Baur D, Hausmann A, Tischer J, Horster S. Anthracycline-induced cardiotoxicity: cardiac monitoring by continuous wave-Doppler ultrasound cardiac output monitoring and correlation to echocardiography. Onkologie. 2012;35(5):241-6. doi: 10.1159/000338335. Epub 2012 Apr 23. PMID 22868502
- [Background] Nguyen HB, Banta DP, Stewart G, Kim T, Bansal R, Anholm J, Wittlake WA, Corbett SW. Cardiac index measurements by transcutaneous Doppler ultrasound and transthoracic echocardiography in adult and pediatric emergency patients. J Clin Monit Comput. 2010 Jun;24(3):237-47. doi: 10.1007/s10877-010-9240-6. Epub 2010 Jun 20. PMID 20563629
- [Background] Van den Oever HL, Murphy EJ, Christie-Taylor GA. USCOM (Ultrasonic Cardiac Output Monitors) lacks agreement with thermodilution cardiac output and transoesophageal echocardiography valve measurements. Anaesth Intensive Care. 2007 Dec;35(6):903-10. doi: 10.1177/0310057X0703500608. PMID 18084981
- [Background] Smith BE, Madigan VM. Non-invasive method for rapid bedside estimation of inotropy: theory and preliminary clinical validation. Br J Anaesth. 2013 Oct;111(4):580-8. doi: 10.1093/bja/aet118. Epub 2013 May 3. PMID 23645929
- See also: Census and Statistics Development, Hong Kong SAR — http://www.censtatd.gov.hk